CLINICAL TRIAL: NCT05808491
Title: Effectiveness of Online Resilience Intervention in Older Adults: A Randomized Clinical Trial
Brief Title: Online Resilience Intervention in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YM108150E
Record Dates: First submitted 2023-03-29; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Health Promotion Program
Keywords: resilience intervention; physical activity; well-being; older adult
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: control group and experimental group
Who Masked: Participant
Masking Description: control group and experimental group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): provide usual care, which includes patient education sheets and medical treatment covered by National Health Insurance regulations
- intervention (Experimental): provide a resilience intervention by teaching participants how to assess their level of resilience and how to minimize their level of stress. Other objectives include to enhance coping, to control belief, and to manage skills through role-play, group discussion, and individual practice.
  Interventions: Radiation: online resilience intervention

INTERVENTIONS:
Radiation: online resilience intervention — online resilience intervention were presented in four 60-minute sections, once a week for four weeks embracing four sections
  Arms: intervention

SUMMARY:
Resilience in older adults is important for Healthy aging. The purpose of this study was to examine the effectiveness of an on-line program of resilience interventions among older adults.

DETAILED DESCRIPTION:
Healthy aging not only free from illness but also need to maintain healthy physical and mental function, be active in social life and contribute to society. Aging bring comprehensive impacts toward family, society and country, especially in individual. Resilience intervention can improve the intrinsic health and well-being for older adults. Good physical activity benefits to healthy aging. The purpose of this study was to examine the effectiveness of an on-line program of resilience interventions among older adults.

ELIGIBILITY:
Inclusion Criteria:

* able to read Chinese, and aged 65 years or older.

Exclusion Criteria:

* with a psychiatric diagnosis and who had a neoplasm

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
the changes from baseline to 1, 3 month of resilience | baseline, 1, 3 month
  measured by The Chinese Version of Resilience Scale
the changes from baseline to 1, 3 month of physical activity | baseline, 1, 3 month
  measured by Physical Activity Scale for the Elderly
the changes from baseline to 1, 3 month of well-being | baseline, 1, 3 month
  measured by well-being scale

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang Ming University, Taipei, Taiwan

REFERENCES:
- [Derived] Wu YC, Shen SF, Chen LK, Tung HH. A Web-Based Resilience-Enhancing Program to Improve Resilience, Physical Activity, and Well-being in Geriatric Population: Randomized Controlled Trial. J Med Internet Res. 2024 Jul 25;26:e53450. doi: 10.2196/53450. PMID 39052335